CLINICAL TRIAL: NCT01061710
Title: Champix Tablets Special Investigation -Retrospective Survey For Subjects Who Have Been Retreated With Champix.-(Regulatory Post Marketing Commitment Plan).
Brief Title: Varenicline (Champix®) Special Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051117
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Smoking Cessation
Keywords: Smoking; smoking cessation; Japanese; varenicline; retreatment; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- varenicline (Champix®): Subjects who have been retreated with varenicline within 52 weeks and have been enrolled to varenicline protocol A3051109.
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: varenicline — Dosage form: tablet 0.5mg, tablet 1mg. The usual adult dosage for oral use is 0.5 mg once daily after eating on Days 1 to 3; 0.5 mg twice daily after eating in the morning and evening on Days 4 to 7, and 1 mg twice daily after eating in the morning and evening on Day 8 and thereafter. The drug should be administered to subjects for 12 weeks.
  Other Names: Chantix, Champix

SUMMARY:
The purpose of this study is to collect the efficacy and safety information in subjects who have been retreated with varenicline (Champix®) within 52 weeks of initial treatment for their appropriate use in daily practice and are participants for varenicline Drug Use Investigation protocol A3051109 ((NCT# NCT00772941).

DETAILED DESCRIPTION:
The subjects have been retreated with varenicline within 52 weeks, and subjects have been enrolled to varenicline Drug Use Investigation protocol A3051109.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects intend to quit tobacco use who are prescribed varenicline (Champix®) by their Physicians
* Subjects who are prescribed varenicline (Champix®) for the second time within 52 weeks of initial treatment.

Exclusion Criteria:

Non-participants of varenicline (Champix®) Drug use Investigation protocol A3051109.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects who have been retreated with varenicline in A3051109 (NCT# NCT00772941) within 52 weeks of initial treatment.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051117&StudyName=Varenicline%20%28Champix%AE%29%20Special%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This survey enrolled those who participated in preceding varenicline Drug Use Investigation protocol A3051109 (NCT00772941) and retreated with varenicline within 52 weeks of initial treatment.
Groups:
- Varenicline (Champix®): The usual adult dosage for oral use is as follows: Day 1 through Day 3, 0.5 mg once daily after eating; Day 4 through Day 7, 0.5 mg twice daily after eating in the morning and evening; and Day 8 and thereafter, 1 mg twice daily after eating in the morning and evening. Treatment period was 12 weeks. Participants were retreated within 52 weeks of initial treatment.
Period: Overall Study
Arm/Group | Varenicline (Champix®)
Started | 20
Completed | 6
Not Completed | 14
Not completed — Protocol Violation | 14

BASELINE CHARACTERISTICS:
Population: A total of 20 participants were enrolled in this survey. Of the 20 participants, 14 participants were excluded from the baseline analysis due to a protocol violation.
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  <65 years | 3
  >=65 years | 3
Sex/Gender, Customized [Number; unit: participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to veranicline in a participant who received veranicline. Treatment related adverse events were evaluated in company with the causal relationship to veranicline.
Time Frame: 24 weeks
Population: The safety analysis population comprised participants who had been enrolled in varenicline protocol A3051109 and retreated with varenicline within 52 weeks of initial treatment.
Measure: Number; unit: Participants
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Responders to Varenicline Treatment
Description: Number of participants who succeeded in smoking cessation from 12 weeks through 24 weeks of the observation period.
Time Frame: 24 weeks
Population: The efficacy analysis population comprised the participants who had at least one post-baseline efficacy measurement among the safety analysis population.
Measure: Number; unit: Participants
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 6
Participants | 2 [4.3 to 77.7]

3. Secondary Outcome: Number of Treatment-Related Adverse Events (AEs) Unlisted in Japanese Package Insert
Description: An AE was any untoward medical occurrence attributed to varenicline in a participant who received varenicline. Treatment related adverse events were evaluated in company with the causal relationship to veranicline.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Number of Participants With Risk Factors Likely to Affect the Frequency of Treatment-Related Adverse Events (AEs)
Time Frame: 24 weeks
Population: The safety analysis population comprised participants who had been enrolled in varenicline protocol A3051109 and retreated with varenicline within 52 weeks of initial treatment. Because of the small population size, no risk analyses were performed.
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Risk Factors Likely to Affect the Proportion of Responders
Time Frame: 24 weeks
Population: The efficacy analysis population comprised the participants who had at least one post-baseline efficacy measurement among the safety analysis population. Because of the small population size, no risk analyses were performed.
Arm/Group | Varenicline (Champix®)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The frequency of adverse events during the survey.
Arm/Group | Varenicline (Champix®)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.